CLINICAL TRIAL: NCT00522873
Title: A Double-blind, Randomized, Multi-center Study to Investigate the Endometrial Safety of a Continuous, Combined, Oral Estrogen/Progestin Preparation (17b-estradiol [E2] / Drospirenone [DRSP]) and to Compare the Bleeding Pattern of Subjects Treated With E2 / DRSP With the Bleeding Pattern of Subjects Treated With E2 / Norethisterone Acetate (NETA) When Used for Hormone Therapy (HT) for 1 Year in Post-menopausal Women
Brief Title: Endometrial Safety Study
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Bayer (Industry)
Collaborators: Laboratorium für Klinische Forschung (Unknown); Diagnostic Cytology Laboratory (Unknown); University of California, San Francisco (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 91508; 2006-006199-39 (EudraCT Number); 310523 (Other: Company internal)
Record Dates: First submitted 2007-08-29; First posted 2007-08-30 (Estimated); Results first posted 2012-06-28 (Estimated); Last update posted 2014-12-31 (Estimated); Status verified 2014-12

CONDITIONS: Postmenopause
Keywords: Postmenopausal Symptoms e.g.; Hot flushes; Sweating episodes; Vaginal dryness
MeSH Terms: conditions — Hot Flashes | interventions — drospirenone; estradiol, norethindrone drug combination

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- 0.25mg DRSP / 0.5mg E2 (BAY86-4891) (Experimental): One capsule [0.25mg drospirenone/0.5mg 17β-estradiol (DRSP/E2)] per day taken orally for 13 cycles (28 days per cycle).
  Interventions: Drug: 0.25mg DRSP / 0.5mg E2 (BAY86-4891)
- 0.5mg NETA / 1.0mg E2 (Activella) (Active Comparator): One capsule [0.5mg norethisterone acetate/1.0mg 17β-estradiol (NETA/E2)] per day taken orally for 13 cycles (28 days per cycle).
  Interventions: Drug: 0.5mg NETA / 1.0mg E2 (Activella)

INTERVENTIONS:
Drug: 0.25mg DRSP / 0.5mg E2 (BAY86-4891) — One capsule [0.25mg drospirenone/0.5mg 17β-estradiol (DRSP/E2)] per day taken orally for 13 cycles (28 days per cycle).
  Arms: 0.25mg DRSP / 0.5mg E2 (BAY86-4891)
Drug: 0.5mg NETA / 1.0mg E2 (Activella) — One capsule [0.5mg norethisterone acetate/1.0mg 17β-estradiol (NETA/E2)] per day taken orally for 13 cycles (28 days per cycle).
  Arms: 0.5mg NETA / 1.0mg E2 (Activella)

SUMMARY:
The study is designed to investigate the safety of the investigational product for the lining of the uterus (endometrium).

ELIGIBILITY:
Inclusion Criteria:

* Postmenopausal women between 40 and 65 years of age with hormone therapy indication (symptoms and need for treatment)
* Non-hysterectomized women.

Exclusion Criteria:

* Usual exclusion criteria for hormone therapy apply.

Ages: 40 Years to 65 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 662 (Actual)
Dates: Start 2007-08; Primary Completion 2009-08 (Actual); Study Completion 2009-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Bayer Study Director, Study Director — Bayer
Locations (51):
- United States (16):
  - Chandler, Arizona
  - San Diego, California
  - Denver, Colorado
  - Greenwood Village, Colorado
  - Boynton Beach, Florida
  - Clearwater, Florida
  - Boise, Idaho
  - Amite, Louisiana
  - Marrero, Louisiana
  - Las Vegas, Nevada
  - Cleveland, Ohio
  - Philadelphia, Pennsylvania
  - Columbia, South Carolina
  - Corpus Christi, Texas
  - Richmond, Virginia
  - Seattle, Washington
- Argentina (3):
  - Lanús Oeste, Buenos Aires
  - San Isidro, Buenos Aires
  - Buenos Aires, Ciudad Auton. de Buenos Aires
- Austria (11):
  - Mödling, Lower Austria
  - Wiener Neustadt, Lower Austria
  - Fürstenfeld, Styria
  - Wörgl, Tyrol
  - Bregenz, Vorarlberg
  - Innsbruck
  - Klagenfurt
  - Mürzzuschlag
  - Sankt Pölten
  - Vienna
  - Zeltweg
- Brazil (4):
  - Goiânia, Goiás
  - Curitiba, Paraná
  - Porto Alegre, Rio Grande do Sul
  - São Paulo, São Paulo
- Denmark (3):
  - Aalborg
  - Ballerup Municipality
  - Vejle
- Italy (8):
  - Bologna
  - Cagliari
  - Modena
  - Novara
  - Parma
  - Pisa
  - Sassari
  - Siena
- Mexico (4):
  - Mexico City, Mexico City
  - México
  - México, D.F.
  - Monterrey
- Russia (2):
  - Moscow
  - Moskva

REFERENCES:
- [Result] Genazzani AR, Schmelter T, Schaefers M, Gerlinger C, Gude K. One-year randomized study of the endometrial safety and bleeding pattern of 0.25 mg drospirenone/0.5 mg 17beta-estradiol in postmenopausal women. Climacteric. 2013 Aug;16(4):490-8. doi: 10.3109/13697137.2013.783797. Epub 2013 May 11. PMID 23531117
- See also: click here and search for Bayer Product information provided by the EMA — http://www.clinicaltrialsregister.eu

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Only non-hysterectomized, postmenopausal women could take part in this study. The women had to have symptoms requiring hormone therapy in the opinion of the investigator. An endometrial biopsy at screening was to show no evidence of endometrial hyperplasia or cancer.
Pre-assignment Details: 944 women screened, 661 treated. 282 failed screening: consent withdrawn (55), in-/exclusion criteria not met (209), lost to follow-up (3), other (15). 1 woman was randomized but not treated (own decision). 5 women completed the study but not study medication, i.e. they stopped medication early but remained in the study for final assessments.
Period: Overall Study
Arm/Group | 0.25mg DRSP / 0.5mg E2 (BAY86-4891) | 0.5mg NETA / 1.0mg E2 (Activella)
Started | 490 | 172
Received Treatment | 489 | 172
Completed | 394 (394 women completed study medication. 398 women completed the study.) | 128 (128 women completed study medication. 129 women completed the study.)
Not Completed | 96 | 44
Not completed — Adverse Event | 41 | 26
Not completed — Withdrawal by Subject | 20 | 9
Not completed — Protocol Violation | 14 | 4
Not completed — Lost to Follow-up | 11 | 3
Not completed — Personal Reasons | 8 | 1
Not completed — Medication Errors | 1 | 1
Not completed — Never Received Medication | 1 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | 0.25mg DRSP / 0.5mg E2 (BAY86-4891) | 0.5mg NETA / 1.0mg E2 (Activella) | Total
Number analyzed (Participants) | 489 | 172 | 661
Age, Continuous [Mean (Standard Deviation); unit: Years] | 53.5 (5.1) | 53.5 (4.5) | 53.5 (4.9)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 489 | 172 | 661
  Male | 0 | 0 | 0
Body Mass Index (BMI) [Mean (Standard Deviation); unit: kg/m^2] — Body mass index was calculated with body weight and height measured at screening (BMI = body weight in kg/ body height in m^2).
  kg/m^2 | 26.315 (4.851) | 26.020 (5.476) | 26.184 (5.008)
Number of participants with hysterectomy/oophorectomy [Number; unit: Participants]
  Hysterectomized | 0 | 0 | 0
  Oophorectomized | 25 | 5 | 30
Years since last menstruation at baseline [Mean (Standard Deviation); unit: years] | 5.109 (4.528) | 4.807 (4.287) | 5.031 (4.465)

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants in the DRSP/E2 Group With an Assessment of Endometrial Hyperplasia or Worse at End of Study (EoS) (1 Year of Treatment)
Description: The number of women who had a biopsy classified as 'hyperplasia or worse' at any time during the study. According to the protocol this endpoint was defined as primary for the DRSP/E2 group only.
Time Frame: Up to one year
Population: For the DRSP/E2 group only - Primary analysis set (PAS): All subjects from the full analysis set (FAS) who either had a biopsy result classified as 'normal' or 'hyperplasia or worse' after a year of treatment or who prematurely discontinued the study before Cycle 13 with a biopsy classified as 'hyperplasia or worse'.
Measure: Number; unit: Participants
Arm/Group | 0.25mg DRSP / 0.5mg E2 (BAY86-4891)
Number analyzed (Participants) | 309
Participants | 0
Statistical Analysis 1: Comparison: 0.25mg DRSP / 0.5mg E2 (BAY86-4891); Exact 95% confidence interval for proportion of participants with hyperplasia or worse at EoS; Test type: Superiority or Other; proportion = 0.0000, 95% CI 2-sided [0.0000 to 0.0119] — The number of women who had a biopsy classified as 'hyperplasia or worse' was divided by the number of women with an evaluable biopsy (i.e. classified as 'normal' after 1 year of treatment or as 'hyperplasia or worse' at any time during the study)

2. Secondary Outcome: Number of Participants With Amenorrhea During Month 1 to 3 of Treatment
Description: The women were to record daily in a diary, indicating 'no bleeding', 'spotting', 'light bleeding', 'normal bleeding' or 'heavy bleeding'. Women were considered to have amenorrhea if they had no bleeding and no spotting day within the given time interval.
Time Frame: Month 1 to Month 3
Population: Per protocol set (PPS): All subjects from the FAS who had at least 75% overall study drug compliance and no major protocol violations
Measure: Number; unit: Participants
Arm/Group | 0.25mg DRSP / 0.5mg E2 (BAY86-4891) | 0.5mg NETA / 1.0mg E2 (Activella)
Number analyzed (Participants) | 371 | 113
Participants | 255 | 67
Statistical Analysis 1: Comparison: 0.25mg DRSP / 0.5mg E2 (BAY86-4891); exact 95% confidence intervall (Clopper-Pearson) for proportion of participants with amenorrhea; Test type: Superiority or Other; proportion = 0.687, 95% CI 2-sided [0.637 to 0.734]
Statistical Analysis 2: Comparison: 0.5mg NETA / 1.0mg E2 (Activella); exact 95% confidence intervall (Clopper-Pearson) for proportion of participants with amenorrhea; Test type: Superiority or Other; proportion = 0.593, 95% CI 2-sided [0.496 to 0.684]

3. Secondary Outcome: Number of Participants With Amenorrhea During Month 10 to 12 of Treatment
Description: The women were to record any bleeding daily in a diary, indicating 'no bleeding', 'spotting', 'light bleeding', 'normal bleeding' or 'heavy bleeding'. Women were considered to have amenorrhea if they had no bleeding and no spotting day within the given time interval.
Time Frame: Month 10 to Month 12
Population: as for outcome 2
Measure: Number; unit: Participants
Arm/Group | 0.25mg DRSP / 0.5mg E2 (BAY86-4891) | 0.5mg NETA / 1.0mg E2 (Activella)
Number analyzed (Participants) | 355 | 106
Participants | 280 | 89
Statistical Analysis 1: Comparison: 0.25mg DRSP / 0.5mg E2 (BAY86-4891); exact 95% confidence intervall (Clopper-Pearson) for proportion of participants with amenorrhea; Test type: Superiority or Other; proportion = 0.789, 95% CI 2-sided [0.743 to 0.830]
Statistical Analysis 2: Comparison: 0.5mg NETA / 1.0mg E2 (Activella); exact 95% confidence intervall (Clopper-Pearson) for proportion of participants with amenorrhea; Test type: Superiority or Other; proportion = 0.840, 95% CI 2-sided [0.756 to 0.904]

ADVERSE EVENTS:
Arm/Group | 0.25mg DRSP / 0.5mg E2 (BAY86-4891) | 0.5mg NETA / 1.0mg E2 (Activella)
Serious Adverse Events (participants affected / at risk) | 16/489 | 6/172
Other Adverse Events (participants affected / at risk) | 172/489 | 63/172
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | 0.25mg DRSP / 0.5mg E2 (BAY86-4891) (N=489) | 0.5mg NETA / 1.0mg E2 (Activella) (N=172)
Lymphadenopathy (Blood and lymphatic system disorders) | 1 | 0
Deafness neurosensory (Ear and labyrinth disorders) | 0 | 1
Hyperparathyroidism (Endocrine disorders) | 0 | 1
Retinal vascular thrombosis (Eye disorders) | 0 | 1
Abdominal pain lower (Gastrointestinal disorders) | 1 | 0
Constipation (Gastrointestinal disorders) | 1 | 0
Faecaloma (Gastrointestinal disorders) | 1 | 0
Large intestinal haemorrhage (Gastrointestinal disorders) | 1 | 0
Pancreatitis acute (Gastrointestinal disorders) | 1 | 0
Cholecystitis (Hepatobiliary disorders) | 1 | 0
Cholelithiasis (Hepatobiliary disorders) | 1 | 0
Appendicitis (Infections and infestations) | 0 | 1
Cellulitis (Infections and infestations) | 1 | 0
Pneumonia (Infections and infestations) | 1 | 0
Splenic rupture (Injury, poisoning and procedural complications) | 1 | 0
Hyperglycaemia (Metabolism and nutrition disorders) | 1 | 0
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 1 | 0
Breast cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Colon adenoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Colon cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Lung neoplasm malignant (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Lymphoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Salivary gland adenoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Carpal tunnel syndrome (Nervous system disorders) | 1 | 0
Grand mal convulsion (Nervous system disorders) | 0 | 1
Transient ischaemic attack (Nervous system disorders) | 1 | 0
Anxiety (Psychiatric disorders) | 1 | 0
Self-injurious ideation (Psychiatric disorders) | 1 | 0
Urinary incontinence (Renal and urinary disorders) | 1 | 0
Asthma (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Hip arthroplasty (Surgical and medical procedures) | 1 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 2% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | 0.25mg DRSP / 0.5mg E2 (BAY86-4891) (N=489) | 0.5mg NETA / 1.0mg E2 (Activella) (N=172)
Abdominal pain (Gastrointestinal disorders) | 6 | 4
Influenza (Infections and infestations) | 21 | 6
Nasopharyngitis (Infections and infestations) | 18 | 2
Urinary tract infection (Infections and infestations) | 9 | 4
Weight increased (Investigations) | 17 | 3
Back pain (Musculoskeletal and connective tissue disorders) | 17 | 2
Pain in extremity (Musculoskeletal and connective tissue disorders) | 12 | 0
Uterine leiomyoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 16 | 4
Headache (Nervous system disorders) | 32 | 7
Depression (Psychiatric disorders) | 9 | 6
Breast pain (Reproductive system and breast disorders) | 21 | 10
Breast tenderness (Reproductive system and breast disorders) | 9 | 5
Cervical dysplasia (Reproductive system and breast disorders) | 11 | 7
Endometrial hypertrophy (Reproductive system and breast disorders) | 13 | 4
Postmenopausal haemorrhage (Reproductive system and breast disorders) | 14 | 9
Hypertension (Vascular disorders) | 15 | 5

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of 60 days or less